CLINICAL TRIAL: NCT01152489
Title: Phase II Study of the Effectiveness of a Device and Distraction for Pediatric Immunization Pain in Multiple Age Groups
Brief Title: A Test of the Effectiveness of a Device and Distraction for Pediatric Immunization Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MMJ Labs LLC (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Amy Baxter MD, MMJ Labs LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H09501; R44HD056647-01A2 (NIH); NCT00910611 (obsolete NCT alias)
Record Dates: First submitted 2010-06-26; First posted 2010-06-29 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Procedural Pain
Keywords: Pain
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care (No Intervention): Immunizations are given with standard care of no pain control
- Experimental (Active Comparator): Vibrating device with cold pack held to arm proximal to injections within the same dermatome; caretakers offered and instructed in use of distraction cards.
  Interventions: Device: Device: Buzzy
- Sham Device (Sham Comparator): The device without batteries or cold pack held to arm proximal to injections. No formal distraction.
  Interventions: Device: Buzzy: sham device

INTERVENTIONS:
Device: Device: Buzzy — "Buzzy", the vibrating cold pack, is held in place with a velcro strap or pressed by caretaker or nurse immediately prior and during immunizations. The vibration is activated and the device remains in place during the shot, moving locations if multiple shots are given. Distraction cards with pictures on one side and questions on the other are shown to the child while the caretaker asks the finding and seeking questions on the back.
  Other Names: Buzzy(R); Flippits(TM)
  Arms: Experimental
Device: Buzzy: sham device — The identical device without batteries or a cold pack is held in place proximal to the site with a velcro strap or pressed by parent or nurse immediately prior to immunizations. The device remains in place throughout the procedure, moving locations to complete multiple shots.
  Other Names: Buzzy
  Arms: Sham Device

SUMMARY:
The hypothesis of this study is that distraction cards used by the caretaker along with a vibrating cold pack placed proximal to the site of immunization will decrease the pain of routine pediatric immunizations when compared to a placebo device or standard care.

DETAILED DESCRIPTION:
Needle pain is the most common and the most feared source of childhood pain, resulting in needle phobia for 10$ of adults. Current standard of care for immunizations in the US is no pain relief. An inexpensive, immediately effective form of needle pain control could reduce needle phobia or vaccine refusal in the long term if demonstrated to be effective for immunization pain.

Distraction can decrease procedural distress in children by 50%. The effect of using a multi-modal pain and distraction relieving approach has not been rigorously studied.

ELIGIBILITY:
Inclusion Criteria:

* children receiving routine immunizations

Exclusion Criteria:

* no caregiver present
* chronic illness requiring frequent injections
* clear cognitive impairments affecting communication

Ages: 4 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pain of immunization | 5 minutes during or immediately after immunizations
  Infants' and toddlers' pain is assessed by coding videotapes using the FLACC (face, legs, activity, crying and consolability) scale. Patients age 4 and older rate pain using self-report via the Faces Pain Scale Revised.

SECONDARY OUTCOMES:
Pain from immunization using observational measures | 5 minutes immediately following immunization
  Caretakers and nurses administering the shots rate pain using a 10cm Visual analog scale from "no pain" to "most pain possible"; duration of infant cry is also assessed following the procedure using coded videotape recordings.
Treatment satisfaction | 5 minutes after immunizations
  10 item scale ranging from "strongly agree" to "strongly disagree" with ten parameters of satisfaction with the methods and concepts of immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Baxter, MD, Principal Investigator — MMJ Labs LLC